CLINICAL TRIAL: NCT06632522
Title: Clinical Study of Radiotherapy Combined With Camrelizumab and Apatinib in the Treatment of Liver Cancer Patients With VP4.
Brief Title: Clinical Study of Radiotherapy Combined With Camrelizumab and Apatinib in the Treatment of Liver Cancer Patients .
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24250-4-02
Record Dates: First submitted 2024-09-05; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Liver Cancer
Keywords: Combined with portal vein tumor thrombus,VP4
MeSH Terms: conditions — Liver Neoplasms | interventions — camrelizumab; apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- radiotherapy combined with Camrelizumab and Apatinib (Experimental): radiotherapy combined with Camrelizumab and Apatinib in the treatment of liver cancer patients with VP4
  Interventions: Drug: radiotherapy combined with Camrelizumab and Apatinib

INTERVENTIONS:
Drug: radiotherapy combined with Camrelizumab and Apatinib — Camrelizumab is administered intravenously (without preventive medication), with a fixed dose of 200mg, with an infusion of 30 min (not less than 20 min and not more than 60 min) every three weeks. Apatinib, 250 mg, taken orally within half an hour after meals, QD, continuously.

SUMMARY:
Clinical study of radiotherapy combined with Camrelizumab and Apatinib in the treatment of liver cancer patients with VP4.

DETAILED DESCRIPTION:
This study is a single-arm, open, prospective and multi-center clinical study, aiming at observing and evaluating the efficacy and safety of radiotherapy combined with Camrelizumab and apatinib in the treatment of patients with VP4 liver cancer.

ELIGIBILITY:
Inclusion Criteria：

1. Patients volunteered to join this study and signed informed consent;
2. ≥18 years old, both men and women;
3. Patients with hepatocellular carcinoma diagnosed by CT/MRI;
4. Clinical liver cancer in Barcelona is stage C with portal vein tumor thrombus (PVTT, VP4), which is not suitable for operation or local treatment, or progresses after operation and/or local treatment;
5. For patients who have progressed after local treatment, local treatment (including but not limited to surgery, hepatic artery embolization, TACE, hepatic artery perfusion, radiofrequency ablation, cryoablation or percutaneous ethanol injection) has been completed at least 4 weeks before the baseline imaging scan, and the toxic reactions caused by local treatment (except alopecia) must be restored to the rating of National Cancer Institute-General Terminology for Adverse Events (NCI-CTCAE v5.0).
6. Never received any systematic treatment for HCC before;
7. Except for tumor thrombus, the number of intrahepatic and extrahepatic lesions is ≤10;
8. The diameter of extrahepatic lesions is ≤ 5 cm;
9. At least one measurable lesion (according to the requirements of RECISTv1.1, the long diameter of the measurable lesion in spiral CT scanning is ≥10 mm or the short diameter of swollen lymph nodes is ≥15 mm; Lesions that have received local treatment in the past (except radiotherapy for target lesions) can be used as target lesions after they are clearly advanced according to RECIST v1.1 standard);
10. Child-Pugh liver function classification is Grade A or Grade B (score ≤7).
11. ECOG score: 0 ~ 1;
12. The expected survival time is ≥12 weeks;
13. The main organ functions meet the following requirements (within 7 days before the start of the study and treatment):

(1) Routine blood examination: (Except hemoglobin, no blood transfusion, no use of granulocyte colony stimulating factor [G-CSF] and no drug correction within 14 days before screening): Absolute neutrophil count ≥1.5×109/L; Platelets ≥50×109/L; Hb ≥90 g/L; (2) Biochemical examination: (albumin was not transfused within 14 days before screening): Serum albumin ≥29 g/L; Serum total bilirubin ≤1.5× upper limit of normal range (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase acidase (AKP)≤5×ULN; Serum creatinine (Cr)≤1.5ULN or Cr clearance rate > 50 mL/min (Cockcroft-Gault formula is as follows).

Male: Cr clearance rate =((140- age) × body weight) /(72× blood Cr) Female: Cr clearance rate =((140- age )× body weight) /(72× blood Cr) × 0.85 body weight unit: kg; Blood Cr unit: mg/mL; (3) The international normalized ratio (INR) is ≤ 2.3 or the prothrombin time (PT) exceeds the range of normal control for ≤6 seconds; (4) Urinary protein < 2+ (if urinary protein ≥2+, 24-hour (h) urinary protein quantification can be performed, and 24-hour urinary protein quantification < 1.0 g can be enrolled).

14. If the patient suffers from active hepatitis B virus (HBV) infection, the HBV- deoxyribonucleic acid (DNA) must be less than 500 IU/mL (if the research center only has a copy/mL detection unit, it must be less than 2500 copy/mL), and he must receive anti-HBV treatment (according to local standard treatment, such as entecavir) for at least 14 days before the start of the research treatment, and he is willing to take the whole course during the research period. Hepatitis C virus (HCV) ribonucleic acid (RNA) positive patients must receive antiviral treatment according to local standard treatment guidelines, and their liver function should be within the level 1 increase of CT CAE.

Fertile women: they must agree to abstain from sex (avoid heterosexual intercourse) or use reliable and effective methods of contraception for at least 120 days from signing the informed consent form until the last administration of the study drug. And the serum HCG test must be negative within 7 days before the start of the study treatment; And must be non-lactating. If a female patient has menstruated, has not yet reached the post-menopausal state (continuous non-menstrual period ≥12 months, and no other reasons have been found except menopause), and has not undergone sterilization surgery (such as hysterectomy, bilateral tubal ligation or bilateral oophorectomy), it is considered that the patient has fertility. For male patients whose partner is a woman of childbearing age, they must agree to abstain from sex for at least 120 days from signing the informed consent form until the last administration of the study drug, or to use reliable and effective methods for contraception. Male subjects must also agree not to donate sperm during the same period. Male subjects whose partners are pregnant must use condoms, and no other contraceptive methods are needed.

Exclusion Criteria：

1. Known hepatobiliary cell carcinoma, sarcomatoid HCC, mixed cell carcinoma and fibreboard cell carcinoma; Have other active malignant tumors except HCC within 5 years or at the same time. Localized tumors that have been cured, such as basal cell carcinoma of skin, squamous cell carcinoma of skin, superficial bladder cancer, prostate cancer in situ, cervical cancer in situ, breast cancer in situ, etc., can be included in the group;
2. The tumor thrombus occupies all the portal vein lumen;
3. Except for tumor thrombus, the number of intrahepatic and extrahepatic lesions is more than 10;
4. The diameter of extrahepatic lesions is more than 5 cm;
5. Patients who are ready to undergo or have previously received organ or allogeneic bone marrow transplantation;
6. Moderate and severe ascites with clinical symptoms (except for those who only show a small amount of ascites on imaging but are not accompanied by clinical symptoms); Uncontrolled or moderate or above pleural effusion and pericardial effusion;
7. Patients who have a history of gastrointestinal bleeding or have a clear tendency of gastrointestinal bleeding within 6 months before the start of the study and treatment, such as: bleeding-risk or severe esophageal and gastric varices, local active gastrointestinal ulcer lesions, and persistent fecal occult blood positive, can not be included in the group (if the fecal occult blood is positive in the baseline period, it can be rechecked, and if it is still positive after the recheck, it needs to undergo gastroduodenoscopy (EGD), and if the EGD indicates bleeding-risk esophageal and gastric varices, it can not be included).
8. Abdominal fistula, gastrointestinal perforation or abdominal abscess occurred within 6 months before the start of the study treatment;
9. Known hereditary or acquired bleeding (such as coagulation dysfunction) or thrombotic tendency, such as hemophilia patients; At present, or in the near future (within 10 days before the start of the study treatment), full-dose oral or injection anticoagulants or thrombolytic drugs have been used for therapeutic purposes (low-dose aspirin and low-molecular-weight heparin are allowed for preventive use);
10. Aspirin (> 325 mg/ day (maximum antiplatelet dose) or dipyridamole, ticlopidine, clopidogrel and cilostazol are currently being used or recently used (within 10 days before the start of the study treatment);
11. Thrombosis or embolism occurred within 6 months before the start of study treatment, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction) and pulmonary embolism;
12. There are clinical symptoms or diseases of the heart that can't be well controlled, such as: (1) according to the standards of new york Heart Association (NYHA) (see Annex 5), the cardiac insufficiency is above grade 5)II or the left ventricular ejection fraction (LVEF) is less than 50%; (2) Unstable angina pectoris; (3) myocardial infarction occurred within one year before the start of study and treatment; (4) Clinically significant supraventricular or ventricular arrhythmia needs treatment or intervention; (5)QTc > 450ms (male); QTc > 470ms (female) (QTc interval is calculated by Fridericia formula; If the QTc is abnormal, it can be continuously tested for three times every 2 minutes, and the average value can be taken);
13. Suffering from high blood pressure, which cannot be well controlled by antihypertensive drugs (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg) (based on the average of BP readings obtained by ≥2 measurements), it is allowed to realize the above parameters by using antihypertensive therapy; Hypertensive crisis or hypertensive encephalopathy has occurred in the past;
14. Major vascular diseases (for example, aortic aneurysm requiring surgical repair or recent peripheral artery thrombosis) occurred within 6 months before the start of study treatment;
15. Severe, unhealed or split wounds and active ulcers or untreated fractures;
16. Received major surgical treatment (except diagnosis) within 4 weeks before the start of the study treatment or expected major surgical treatment during the study period;
17. Can't swallow pills, malabsorption syndrome or any condition that affects gastrointestinal absorption;
18. Have suffered from intestinal obstruction and/or clinical signs or symptoms of gastrointestinal obstruction within 6 months before starting the study and treatment, including incomplete obstruction related to the original disease or requiring routine parenteral hydration, parenteral nutrition or tube feeding:
19. At the initial diagnosis, patients with incomplete obstruction/obstruction syndrome/signs/symptoms of intestinal obstruction may be enrolled in the study if they receive definite (surgical) treatment to relieve symptoms;
20. There is evidence that there is pneumoperitoneum that cannot be explained by puncture or recent surgical operation;
21. Past or present central nervous system metastasis;
22. Metastatic diseases involving major airways or blood vessels (for example, portal vein trunk or vena cava that is completely occluded due to tumor invasion needs to be excluded, portal vein trunk refers to the confluence of splenic vein and superior mesenteric vein and the branch where hepatic portal vein divides into left and right branches) or large mediastinal tumor mass in the center (< 30 mm from carina);
23. Those with a history of hepatic encephalopathy;
24. At present, patients with interstitial pneumonia or interstitial lung disease, or patients with previous history of interstitial pneumonia or interstitial lung disease requiring hormone therapy, or other subjects with pulmonary fibrosis, organized pneumonia (for example, bronchiolitis obliterans), pneumoconiosis, drug-related pneumonia, idiopathic pneumonia, or subjects with evidence of active pneumonia or severe impairment of lung function on chest computed tomography (CT) during screening period are allowed to have radiation fields. Active tuberculosis;
25. Active autoimmune disease or history of autoimmune disease and possible recurrence (including but not limited to autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism [subjects who can only be controlled by hormone replacement therapy can be included]); Subjects suffering from skin diseases without systematic treatment, such as vitiligo, psoriasis, alopecia, controlled type I diabetes treated with insulin or asthma in childhood have been completely relieved, and adults can be included without any intervention; Asthmatic patients who need bronchodilators for medical intervention cannot be included;
26. Use immunosuppressant or systemic hormone therapy within 14 days before starting the study treatment to achieve the purpose of immunosuppression (dosage > 10mg/ day of prednisone or other therapeutic hormones);
27. Strong CYP3A4/ CYP2C19 inducers used within 14 days before starting the study treatment include rifampicin (and its analogues) and Hypericum perforatum or strong CYP3A4/ CYP2C19 inhibitors;
28. It is known that there is a serious allergic history to any monoclonal antibody and anti-angiogenesis targeted drugs;
29. Severe infection within 4 weeks before the start of study treatment, including but not limited to hospitalization due to infection, bacteremia or complications of severe pneumonia; Therapeutic antibiotics were given orally or intravenously within 2 weeks before the start of the study treatment (patients receiving preventive antibiotics (for example, patients who prevent urinary tract infection or exacerbation of chronic obstructive pulmonary disease are eligible to participate in the study); 30 patients with congenital or acquired immune deficiency (such as HIV infection);

31. Co-infection with hepatitis B and hepatitis C; 32. Previously received other anti-PD-1 antibody therapy or other immunotherapy against PD-1/PD-L1, or previously received apatinib and sorafenib therapy; 33. Palliative radiotherapy for non-target lesions allowed to control symptoms must be completed at least 2 weeks before the start of the study treatment, and the adverse events caused by radiotherapy have not recovered to ≤ CTCAE level 1; 34. Received live attenuated vaccine treatment within 28 days before the start of the study treatment, or expected to be vaccinated during the treatment period of Karelizumab or within 60 days after the last dose of Karelizumab; 35. Have received other experimental drugs within 28 days before starting the study treatment; According to the researcher's judgment, the patient has other factors that may affect the research results or lead to the forced termination of this study, such as alcoholism, drug abuse, other serious diseases (including mental illness) that need to be treated together, serious laboratory abnormalities, family or social factors, which will affect the safety of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-10-20 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival | up to 3 years
  The time from the beginning of treatment to the progression of the disease or death from any cause.

SECONDARY OUTCOMES:
Progression-free survival | up to 3 years
  Time elapsed from treatment to death from any cause
Objective response rate | up to 3 years
  The proportion of patients with a confirmed complete response or partial response
Disease control rate | up to 3 years
  The proportion of patients who have achieved complete remission (CR), partial remission (PR) or disease stability (SD) at least once after receiving the treatment of this research scheme.

CONTACTS AND LOCATIONS:
Overall Officials: Gong Li, M.A., Study Director — Tsinghua Chang Gung Hospital
Locations (1):
- Beijing Tsinghua Chang Gung Hospital, Beijing, Beijing Municipality, China